CLINICAL TRIAL: NCT04386668
Title: Let It Out (LIO) and COVID19: a Randomised Controlled Trial of an Online Emotional Disclosure-based Intervention for Adults During the COVID19 Pandemic
Brief Title: Let It Out (LIO) and COVID19: Testing an Online Emotional Disclosure-based Intervention During the COVID19 Pandemic
Acronym: LIO-C
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis indicated adaptations to intervention may be required.
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 15281/003
Record Dates: First submitted 2020-05-12; First posted 2020-05-13 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: COVID19
Keywords: COVID19; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIO-C (Experimental): Participants receive LIO-C writing intervention
  Interventions: Other: Let It Out (LIO)-C
- Neutral writing control (Placebo Comparator): Participants receive neutral writing control intervention
  Interventions: Other: Neutral writing control

INTERVENTIONS:
Other: Let It Out (LIO)-C — Participants complete three online 20-minute writing sessions in response to prompts asking them to write about their experiences during the COVID19 pandemic from a self-compassionate perspective
  Other Names: expressive writing; emotional disclosure; expressive disclosure; therapeutic writing
  Arms: LIO-C
Other: Neutral writing control — Participants complete three online 20-minute writing sessions in response to neutral writing prompts
  Arms: Neutral writing control

SUMMARY:
A randomised controlled trial designed to test whether an online expressive writing intervention (LIO-C) can reduce distress for English-speaking adults during the global COVID19 pandemic.

Hypothesis: LIO-C will improve distress (as measured by K10) in adults at 1 week post-intervention compared to a neutral writing control during the COVID19 pandemic.

DETAILED DESCRIPTION:
The world is currently experiencing unprecedented challenges caused by the global coronavirus (COVID19) pandemic. Many countries are enforcing measures to restrict movement of people to reduce the spread of the outbreak, including lock-downs, social distancing and self-isolation. These methods, although necessary to slow the spread of disease, will have negative effects on psychological well-being of large populations. Shortage of health care professionals and measures to restrict interpersonal contact means facilitated psychological interventions will not be feasible for many, at least during the height of the pandemic. There is therefore a need for self-directed psychological interventions that can be practically and quickly implemented online.

Emotional disclosure-based therapies, such as expressive writing (EW), hold potential as low-cost, easy to implement means of support, with minimal requirement for facilitation. In its original format, EW involved writing daily for 15-20 minutes for 3-4 days about a traumatic event. Since its development, it has been adapted in many ways, including writing about positive events and writing about stress from a compassionate stance. There is evidence that such interventions can provide significant psychological and physical benefits in healthy populations and reduce the effects of natural disasters on health and well-being. However, to our knowledge this form of psychological intervention has not been tested during a rapidly evolving crisis or pandemic.

The aim of this study is to test whether an online self-compassion and EW based intervention (LIO-C) can reduce the negative effects of the COVID19 pandemic on health and well-being. The intervention is based on an existing intervention, LIO, that we previously developed for use in advanced disease populations, in collaboration with clinical and health psychologists, and patient and public representatives. For this study, we have adapted the intervention for people living through the current COVID19 pandemic by altering the writing prompts, and translating the intervention to an online hub. As this is an unfacilitated intervention, the instructions involve writing from a compassionate stance to minimise any potential short term negative effects associated with writing about difficult experiences.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults over the age of 18
* Able to read and write clearly in English

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2020-07-12 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Kessler Psychological Distress Scale (K10) | 1 week post-intervention
  10-item self-report distress scale

SECONDARY OUTCOMES:
Kessler Psychological Distress Scale (K10) | Immediately and 8 weeks post-intervention
  10-item self-report distress scale
Perceived Stress Scale (PSS-10) | Immediately, 1 week and 8 weeks post-intervention
  Self-report stress scale
Pittsburgh Sleep Quality Index (PSQI) | Immediately, 1 week and 8 weeks post-intervention
  Self-report sleep scale
Self-compassion scale (SCS) | Immediately, 1 week and 8 weeks post-intervention
  Self-report self-compassion scale
UCLA Loneliness Scale (UCLA LS) | Immediately, 1 week and 8 weeks post-intervention
  Self-report loneliness scale
Uptake of existing mental health services (MHS) | Immediately, 1 week and 8 weeks post-intervention
  Self-report measure of MHS usage
Mood and meaning | Immediately after each writing session
  3-item, 7-point, Likert scale measuring how personal and meaningful participants' felt their writing was and their mood
Acceptability | Immediately post-intervention
  Via an online feedback form

CONTACTS AND LOCATIONS:
Overall Officials: Nuriye Kupeli, Principal Investigator — Marie Curie Palliative Care Research Department, UCL
Locations (1):
- University College London, London, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Fully anonymised participant data will be made available open access via ESRC data repository ReShare
Access Criteria: Open access